CLINICAL TRIAL: NCT04648644
Title: Application of ERAS Protocol in Emergency Surgery
Acronym: ERAS in CDU
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: ERAS in CDU
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Enhanced Recovery After Surgery; Emergency Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: All patients undergoing emergency abdominal surgery for infection or occlusion and treated with bowel resection with or without anastomosis; intestinal bypass or adhesiolysis
  Interventions: Other: Application of ERAS protocol

INTERVENTIONS:
Other: Application of ERAS protocol — Application of a standardized ERAS protocol for the perioperative perioperative management of patients undergoing emergency surgery

SUMMARY:
This study defines a standardized protocol inspired to the ERAS philosophy for the peri-operative treatment of patients undergoing emergency abdominal surgery. Primary endpoint is the feasibility of the application of the standardized protocol; secondary endpoint is the safety

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing emergency abdominal surgery for abdominal sepsis or occlusion and treated with bowel resection with or without anastomosis, intestinal bypass or adhesiolysis.

Exclusion Criteria:

* age <18
* emergency surgery for post-operative complications of post diagnostic procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing emergency surgery for abdominal sepsis or occlusion and treated with bowel resection with or without anastomosis, intestinal bypass or adhesiolysis.
Sampling Method: Non-Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility: % of application of post-operative ERAS items | 30 days
  Compliance to the standardize protocol for each item

SECONDARY OUTCOMES:
Safety: complications rate within 30 days | 30 days
  Complication rate and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Marco Braga, MD, Principal Investigator — University of Milano Bicocca
Locations (8):
- Italy (8):
  - Ospedale Manzoni, Lecco, LC
  - ASST Monza, Monza, MB
  - Ospedale San Raffaele, Milan, Mi
  - ASST Lodi, Lodi
  - Azienda ospedaliero-universitaria Pisana,Ospedale Cisanello, Pisa
  - Ospedale San Jacopo, Pistoia
  - Policlinico Gemelli, Roma
  - Ospedale di Cattinara, Trieste

IPD SHARING:
Plan to Share IPD: No